CLINICAL TRIAL: NCT01785238
Title: Renal Prognosis of Former Preterm Infants 3 to 10 Years After Neonatal Acute Renal Failure
Brief Title: Nephronic Reduction After Neonatal Acute Renal Failure in Preterm
Acronym: IRENEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC12_0238
Record Dates: First submitted 2013-01-18; First posted 2013-02-07 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Neonatal Acute Renal Failure in Preterm
Keywords: preterm infants; acute renal failure; nephronic reduction
MeSH Terms: conditions — Acute Kidney Injury | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cases with neonatal acute renal failure in preterm (Experimental)
  Interventions: Other: renal echography; Other: Blood sampling; Other: collection of an urine sample; Other: Blood pressure measurement
- controls without neonatal acute renal failure in preterm (Other)
  Interventions: Other: renal echography; Other: Blood sampling; Other: collection of an urine sample; Other: Blood pressure measurement

INTERVENTIONS:
Other: renal echography — renal echography to analyse the kidney
Other: Blood sampling — Blood sampling to analyse different parameters of renal function
Other: collection of an urine sample — Collection of an urine sample to perform analysis of renal function parameters
Other: Blood pressure measurement

SUMMARY:
The aim of this study is to evaluate the signs of nephronic reduction in preterm infants who have presented neonatal acute renal failure. The investigators hypothesize that signs of nephronic reduction would appear earlier in former preterm with neonatal acute renal failure than in control preterm infants.

DETAILED DESCRIPTION:
50 former preterm infants who presented acute renal failure will be evaluated between 3 to 10 years.

They will be compared to 25 control former preterm infants without renal dysfunction for signs of nephronic reduction.

At inclusion, in order to analyse renal function, all infants will have blood sampling, renal echography and blood pressure measurement. Urine sample will also be collected.

Two months later, parents will be informed on the results.

ELIGIBILITY:
Inclusion Criteria:

* For both group of cases (50 infants having presented acute renal failure in preterm) AND group of control cases (25 infants without this) :former preterm infant born before 33 weeks of gestational age between january 2003 and june 2010 and hospitalized in the neonatal intensive care unit of Nantes University Hospital.
* Specific to cases: neonatal acute renal failure: serum creatinine>130 micromol/l from the third day of life.
* Control cases: no such renal dysfunction

Exclusion Criteria:

* no parental consent
* other causes of renal failure: congenital uropathy, congenital nephropathy
* congenital cardiopathy, polymalformative syndrome

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
microalbuminuria | Day 1 (at inclusion)
  The primary outcome of this study is to prove that former preterm infants with neonatal acute renal failure are at higher risk of nephronic reduction than control former preterm infants and that they will present microalbuminuria as earlier sign of nephronic reduction. Precisely, if microalbuminuria divided by creatinuria is above 20mg/g or 2mg/mmol, it will be considered as pathologic.

SECONDARY OUTCOMES:
measurement of blood pressure | Day 1 (at inclusion)
  Evaluation of other renal parameters: blood pressure, renal filtration, tubular functions evaluation of renal size and differentiation by ultrasound
measurement of length and volume of kidney by renal echography | day 1
creatinine clearance | day 1
calciuria | Day 1
sodium clearance | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Emma ALLAIN-LAUNAY, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU of Nantes, Nantes, France

REFERENCES:
- [Derived] Bruel A, Roze JC, Quere MP, Flamant C, Boivin M, Roussey-Kesler G, Allain-Launay E. Renal outcome in children born preterm with neonatal acute renal failure: IRENEO-a prospective controlled study. Pediatr Nephrol. 2016 Dec;31(12):2365-2373. doi: 10.1007/s00467-016-3444-z. Epub 2016 Jun 22. PMID 27335060